CLINICAL TRIAL: NCT01265732
Title: An Open Label, Randomized 3-Way Crossover Single Dose Study To Compare The Pharmacokinetics And Relative Bioavailability Of PF-04191834 Using An Oral Wet-Milled Suspension Formulation Versus An Oral Single Dose Dispersion Formulation Under Fasted Conditions In Healthy Volunteers
Brief Title: A Comparison Of The Pharmacokinetics Of PF-04191834 Following Single Dose Administration Of A Dispersion Formulation And A Suspension Formulation In Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0041012
Record Dates: First submitted 2010-11-30; First posted 2010-12-23 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Phase 1; relative bioavailability; healthy volunteers; pharmacokinetics; suspension; dispersion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- oral single dose dispersion 100mg (Active Comparator): Subjects receive a single dose of PF-04191834 as a dispersion
  Interventions: Drug: PF-04191834
- oral wet milled suspension 100mg (Active Comparator): Subjects receive a single dose of PF-04191834 as a suspension
  Interventions: Drug: PF-04191834
- oral wet milled suspension 300mg (Active Comparator): Subjects receive a single dose of PF-04191834 as a suspension
  Interventions: Drug: PF-04191834

INTERVENTIONS:
Drug: PF-04191834 — single dose, 100mg, dispersion
  Arms: oral single dose dispersion 100mg
Drug: PF-04191834 — single dose, 100mg, suspension
  Arms: oral wet milled suspension 100mg
Drug: PF-04191834 — single dose, 300mg, suspension
  Arms: oral wet milled suspension 300mg

SUMMARY:
This study investigates the safety, tolerability and pharmacokinetics of PF-04191834 when respectively given orally as a single dispersion dose and a single dose of a suspension. The suspension is the test formulation and the dispersion is the formulation with which the novel preparation will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg(110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinical evidence of existing hepatic disease or a medical history of such a condition in the last year. Subjects with AST or ALT >ULN. Subjects with total bilirubin >ULN (except those with a documented history of Gilbert's Syndrome). Subjects with AST/ALT/total bilirubin >ULN and <1.5X ULN may be retested once.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication;
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day;
* Females of childbearing potential.
* Subjects with positive responses (score 1) for suicidality on the Sheehan Suicidality Tracking Scale (S-STS) (specifically items 1a, 1b, 3, 4, 5, 6, 7, or 9).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Time of maximum concentration(Tmax) of PF-04191834 in plasma. | 3 days
Area under the curve (AUClast) from the time of dosing to the last data point taken for PF-04191834. | 3 days
Area under the curve from the time of dosing extrapolated to infinity(AUCinf) of PF-04191834. | 3 days

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for PF-04191834 in plasma. | 3 days
Elimination half-life (t1/2) of PF-04191834 | 3 days
Sheehan suicidality tracking scale (SSTS) | Screening and last Day of Period 3
Number of adverse events in patients as a measure of safety and tolerability. | Throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0041012&StudyName=A%20Comparison%20Of%20The%20Pharmacokinetics%20Of%20PF-04191834%20Following%20Single%20Dose%20Administration%20Of%20A%20Dispersion%20Formulation%20And%20A%20Suspension%20Form